CLINICAL TRIAL: NCT01747447
Title: VITamin D and OmegA-3 TriaL: Effects on Bone Structure and Architecture
Brief Title: VITamin D and OmegA-3 TriaL: Effects on Bone Structure and Architecture (VITAL)
Acronym: VITAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Meryl LeBoff, Director of Skeletal Health and Osteoporosis Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012P000560; 1R01AR059775-01A1 (NIH); 5R01AR060574-03 (NIH)
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Results first posted 2021-03-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Bone Density; Body Composition; Bone Health
MeSH Terms: interventions — Fatty Acids, Omega-3; Fish Oils; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D placebo + fish oil placebo (Placebo Comparator): Daily vitamin D placebo and daily fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 placebo; Dietary Supplement: Fish oil placebo
- Vitamin D placebo + fish oil (Active Comparator): Daily vitamin D placebo and daily fish oil capsule (1 g/d; EPA + DHA in a 1.2:1 ratio)
  Interventions: Dietary Supplement: Vitamin D3 placebo; Dietary Supplement: omega-3 fatty acids (fish oil)
- Vitamin D + fish oil placebo (Active Comparator): Daily vitamin D (2,000 IU/d) and daily fish oil placebo
  Interventions: Dietary Supplement: Fish oil placebo; Dietary Supplement: Vitamin D3
- Vitamin D + fish oil (Active Comparator): Daily vitamin D (2,000 IU/d) and daily fish oil capsule (1 g/d; EPA + DHA in a 1.2:1 ratio)
  Interventions: Dietary Supplement: omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 placebo — Vitamin D placebo
  Arms: Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo
Dietary Supplement: Fish oil placebo — Fish oil placebo
  Arms: Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo
Dietary Supplement: omega-3 fatty acids (fish oil) — Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil
Dietary Supplement: Vitamin D3 — Vitamin D3 (cholecalciferol), 2000 IU per day.
  Other Names: cholecalciferol
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is a randomized clinical trial in 25,871 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or fish oil (1 gram of omega-3 fatty acids) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among a sub-cohort of 771 participants in VITAL and will test the efficacy and safety of high-dose vitamin D supplementation vs. placebo on skeletal health and body composition.

DETAILED DESCRIPTION:
The VITAL: Effects on Bone Structure and Architecture is an ancillary study of the parent VITAL. This study has enrolled a sub-cohort of 771 VITAL participants at the NIH-sponsored Harvard Catalyst Clinical and Translational Science Center (CTSC). The following measurements will be performed at baseline and 2 years post-randomization to determine whether high-dose vitamin D supplementation vs. placebo: 1) produces small increases or reduces bone loss in spine, hip, and total body areal bone density as assessed by dual x-ray absorptiometry (DXA); 2) reduces bone turnover as assessed by biomarkers of bone resorption and formation; 3) improves (a) volumetric bone mineral density (vBMD) and measures of bone structure as assessed by peripheral quantitative computed tomography (pQCT) and (b) bone microarchitecture as assessed by high resolution pQCT (HR-pQCT) at the distal radius and tibia as well as trabecular bone score (TBS) at the spine; and 4) results in changes in body composition as assessed by DXA. Parallel assessments of the effects of omega-3 fatty acids will be performed. This study may elucidate the mechanisms through which high-dose vitamin D may prevent age-related fractures and provide new insights into the role of vitamin D on skeletal health and body composition.

We are currently analyzing the effects of daily dietary supplements of fish oil (1 gram of omega-3 fatty acids) vs. placebo on skeletal health and body composition.

ELIGIBILITY:
Participants in VITAL (NCT 01169259) who meet the following criteria are eligible to participate in this ancillary study:

* Those who are using bisphosphonates currently or within the past 2 years, or other bone-active medications currently or within the past year are not eligible for this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 771 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meryl S LeBoff, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] LeBoff MS, Yue AY, Copeland T, Cook NR, Buring JE, Manson JE. VITAL-Bone Health: rationale and design of two ancillary studies evaluating the effects of vitamin D and/or omega-3 fatty acid supplements on incident fractures and bone health outcomes in the VITamin D and OmegA-3 TriaL (VITAL). Contemp Clin Trials. 2015 Mar;41:259-68. doi: 10.1016/j.cct.2015.01.007. Epub 2015 Jan 24. PMID 25623291
- [Background] Donlon CM, LeBoff MS, Chou SH, Cook NR, Copeland T, Buring JE, Bubes V, Kotler G, Manson JE. Baseline characteristics of participants in the VITamin D and OmegA-3 TriaL (VITAL): Effects on Bone Structure and Architecture. Contemp Clin Trials. 2018 Apr;67:56-67. doi: 10.1016/j.cct.2018.02.003. Epub 2018 Feb 23. PMID 29408561
- [Background] Goldman AL, Donlon CM, Cook NR, Manson JE, Buring JE, Copeland T, Yu CY, LeBoff MS. VITamin D and OmegA-3 TriaL (VITAL) bone health ancillary study: clinical factors associated with trabecular bone score in women and men. Osteoporos Int. 2018 Nov;29(11):2505-2515. doi: 10.1007/s00198-018-4633-3. Epub 2018 Jul 18. PMID 30022253
- [Background] LeBoff MS, Chou SH, Murata EM, Donlon CM, Cook NR, Mora S, Lee IM, Kotler G, Bubes V, Buring JE, Manson JE. Effects of Supplemental Vitamin D on Bone Health Outcomes in Women and Men in the VITamin D and OmegA-3 TriaL (VITAL). J Bone Miner Res. 2020 May;35(5):883-893. doi: 10.1002/jbmr.3958. Epub 2020 Jan 30. PMID 31923341
- [Derived] Chou SH, Murata EM, Yu C, Danik J, Kotler G, Cook NR, Bubes V, Mora S, Chandler PD, Tobias DK, Copeland T, Buring JE, Manson JE, LeBoff MS. Effects of Vitamin D3 Supplementation on Body Composition in the VITamin D and OmegA-3 TriaL (VITAL). J Clin Endocrinol Metab. 2021 Apr 23;106(5):1377-1388. doi: 10.1210/clinem/dgaa981. PMID 33513226
- [Derived] LeBoff MS, Murata EM, Cook NR, Cawthon P, Chou SH, Kotler G, Bubes V, Buring JE, Manson JE. VITamin D and OmegA-3 TriaL (VITAL): Effects of Vitamin D Supplements on Risk of Falls in the US Population. J Clin Endocrinol Metab. 2020 Sep 1;105(9):2929-38. doi: 10.1210/clinem/dgaa311. PMID 32492153
- See also: VITAL Study Website — http://www.vitalstudy.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The data were presented as Active Vitamin D + Active Omega-3 fatty acids, Active Vitamin D + Placebo Omega-3 fatty acids, Placebo Vitamin D + Active Omega-3 fatty acids, and Placebo Vitamin D + Placebo Omega-3 fatty acids.
Groups:
- ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids: Received active Vitamin D and active omega-3 fatty acids
- ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids: Received active Vitamin D and placebo omega-3 fatty acids
- PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids: Received placebo Vitamin D and active omega-3 fatty acids
- PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids: Received placebo Vitamin D and placebo omega-3 fatty acids
Period: Overall Study
Arm/Group | ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids | ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids | PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids | PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids
Started | 193 | 195 | 195 | 188
Completed | 170 | 177 | 176 | 164
Not Completed | 23 | 18 | 19 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids | ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids | PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids | PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids | Total
Number analyzed (Participants) | 193 | 195 | 195 | 188 | 771
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 119 | 117 | 118 | 112 | 466
  >=65 years | 74 | 78 | 77 | 76 | 305
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (6.5) | 63.7 (5.5) | 64 (6.3) | 63.9 (6.3) | 63.8 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 91 | 97 | 84 | 360
  Male | 105 | 104 | 98 | 104 | 411
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 3 | 6 | 10 | 29
  Not Hispanic or Latino | 172 | 183 | 179 | 169 | 703
  Unknown or Not Reported | 11 | 9 | 10 | 9 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Of the total 771 participants, only 755 participants self-reported their race & ethnic group.
  Participants
    number analyzed (Participants) | 190 | 193 | 189 | 183 | 755
    Non-Hispanic White | 155 | 162 | 157 | 156 | 630
    African American | 18 | 17 | 17 | 15 | 67
    Hispanic (non-African American) | 8 | 3 | 6 | 9 | 26
    Asian/Pacific Islander | 5 | 4 | 4 | 2 | 15
    American Indian/Alaskan Native | 1 | 1 | 3 | 0 | 5
    Other | 3 | 6 | 2 | 1 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 193 | 195 | 195 | 188 | 771
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (4.7) | 26.9 (4.7) | 27.7 (5.0) | 26.8 (4.6) | 27.2 (4.8)
Fat Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 10.3 (4.1) | 10.2 (3.9) | 10.7 (3.8) | 9.9 (3.6) | 10.3 (3.9)
Leisure Time Physical Activity [Median (Inter-Quartile Range); unit: hr/wk] | 22.7 [9.7 to 43.7] | 21.5 [7.7 to 35.6] | 21.6 [8.4 to 36.0] | 20.4 [6.9 to 36.9] | 21.5 [6.9 to 43.7]
Diabetes History [Count of Participants; unit: Participants] | 20 | 24 | 18 | 21 | 83
Current Smoking [Count of Participants; unit: Participants] | 14 | 12 | 9 | 13 | 48
Any Fracture History [Count of Participants; unit: Participants] | 13 | 19 | 15 | 14 | 61
Parental History of Hip Fracture [Count of Participants; unit: Participants] | 23 | 31 | 24 | 24 | 102
Baseline Calcium Supplement Use [Count of Participants; unit: Participants] | 29 | 40 | 36 | 27 | 132
Baseline Vitamin D Use [Count of Participants; unit: Participants] | 70 | 87 | 92 | 77 | 326
Baseline Total 25(OH)D [Mean (Standard Deviation); unit: ng/mL] | 27.1 (8.5) | 26.9 (9.2) | 28.9 (10.1) | 28.0 (8.5) | 27.7 (9.1)
Baseline Free 25(OH)D [Mean (Standard Deviation); unit: pg/mL] | 5.9 (1.8) | 5.6 (1.8) | 6.0 (2.1) | 5.8 (1.7) | 5.8 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Density
Description: To determine whether vitamin D and/or omega-3 supplementation produces small increases or reduces bone loss in spine, hip, and total body areal bone density, as assessed by DXA. Reported values are rounded up.
Time Frame: 2 years
Population: Some measurements were excluded due to metal artifacts, severe osteoarthritis, severe scoliosis, degenerative disc disease, and bilateral breast implants.
Measure: Mean (Standard Deviation); unit: g/cm^2
Groups:
- Active Vitamin D: Received active Vitamin D
- Vitamin D Placebo: Received placebo Vitamin D
- Active Omega-3 Fatty Acids: Received active omega-3 fatty acids
- Omega-3 Fatty Acids Placebo: Received placebo omega-3 fatty acids
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 388 | 383 | 388 | 383
g/cm^2
  Baseline Spine Areal Bone Mineral Density: number analyzed (Participants) | 368 | 352 | 359 | 361
  Baseline Spine Areal Bone Mineral Density | 1.02 (0.16) | 1.02 (0.17) | 1.02 (0.16) | 1.02 (0.17)
  Year 2 Spine Areal Bone Mineral Density: number analyzed (Participants) | 327 | 307 | 315 | 319
  Year 2 Spine Areal Bone Mineral Density | 1.03 (0.16) | 1.03 (0.17) | 1.03 (0.17) | 1.03 (0.17)
  Baseline Femoral Neck Hip Areal Bone Mineral Density: number analyzed (Participants) | 380 | 381 | 385 | 376
  Baseline Femoral Neck Hip Areal Bone Mineral Density | 0.77 (0.13) | 0.77 (0.13) | 0.77 (0.13) | 0.76 (0.12)
  Year 2 Femoral Neck Hip Areal Bone Mineral Density: number analyzed (Participants) | 336 | 339 | 342 | 333
  Year 2 Femoral Neck Hip Areal Bone Mineral Density | 0.77 (0.13) | 0.77 (0.12) | 0.77 (0.13) | 0.76 (0.12)
  Baseline Total Hip Areal Bone Mineral Density: number analyzed (Participants) | 384 | 381 | 386 | 379
  Baseline Total Hip Areal Bone Mineral Density | 0.94 (0.15) | 0.93 (0.15) | 0.94 (0.15) | 0.93 (0.15)
  Year 2 Total Hip Areal Bone Mineral Density: number analyzed (Participants) | 340 | 339 | 343 | 336
  Year 2 Total Hip Areal Bone Mineral Density | 0.93 (0.15) | 0.94 (0.15) | 0.94 (0.15) | 0.93 (0.15)
  Baseline Whole Body Areal Bone Mineral Density: number analyzed (Participants) | 371 | 369 | 373 | 367
  Baseline Whole Body Areal Bone Mineral Density | 1.15 (0.13) | 1.15 (0.13) | 1.15 (0.13) | 1.15 (0.13)
  Year 2 Whole Body Areal Bone Mineral Density: number analyzed (Participants) | 310 | 318 | 317 | 311
  Year 2 Whole Body Areal Bone Mineral Density | 1.15 (0.13) | 1.15 (0.13) | 1.15 (0.13) | 1.15 (0.13)

2. Primary Outcome: Bone Turnover P1NP
Description: To determine whether vitamin D and/or omega-3 supplementation reduces bone turnover, assessed biomarkers of bone formation (propeptide of type 1 collagen [P1NP]).
Time Frame: 2 years
Population: The original lab performing the assays for the bone turnover markers closed. Thus, the assays were payed for using divisional funds, resulting in a decrease in the total number of samples analyzed. The analysis population was a representative sample of the overall cohort.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 200 | 200 | 205 | 195
ug/L
  Baseline P1NP | 49.99 (19.70) | 49.29 (19.47) | 50.25 (20.83) | 48.99 (18.18)
  Year 2 P1NP | 48.28 (16.74) | 49.04 (18.42) | 48.00 (18.69) | 49.36 (16.35)

3. Secondary Outcome: Change in Bone Structure
Description: To determine whether vitamin D and/or omega-3 supplementation results in changes in bone structure.
Time Frame: 2 years
Population: Some participants excluded due to motion
Measure: Mean (Standard Deviation); unit: mg/cm^3
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 388 | 383 | 388 | 383
mg/cm^3
  Baseline Total Volumetric Bone Mineral Density at the Radius: number analyzed (Participants) | 326 | 321 | 330 | 317
  Baseline Total Volumetric Bone Mineral Density at the Radius | 369.68 (69.48) | 373.90 (72.50) | 371.28 (68.72) | 372.29 (73.35)
  Year 2 Total Volumetric Bone Mineral Density at the Radius: number analyzed (Participants) | 282 | 278 | 291 | 269
  Year 2 Total Volumetric Bone Mineral Density at the Radius | 376.24 (74.48) | 382.25 (71.68) | 377.60 (70.42) | 380.98 (75.98)
  Baseline Trabecular Volumetric Bone Mineral Density at the Radius: number analyzed (Participants) | 326 | 321 | 330 | 317
  Baseline Trabecular Volumetric Bone Mineral Density at the Radius | 196.45 (43.16) | 202.80 (46.07) | 197.50 (46.07) | 201.78 (43.20)
  Year 2 Trabecular Volumetric Bone Mineral Density at the Radius: number analyzed (Participants) | 282 | 278 | 291 | 269
  Year 2 Trabecular Volumetric Bone Mineral Density at the Radius | 199.56 (44.65) | 205.11 (46.02) | 200.12 (47.72) | 204.69 (42.67)
  Baseline Cortical Volumetric Bone Mineral Density at the Radius: number analyzed (Participants) | 311 | 308 | 317 | 302
  Baseline Cortical Volumetric Bone Mineral Density at the Radius | 1197.75 (31.57) | 1196.98 (30.82) | 1197.87 (31.45) | 1196.85 (30.93)
  Year 2 Cortical Volumetric Bone Mineral Density at the Radius: number analyzed (Participants) | 258 | 257 | 273 | 242
  Year 2 Cortical Volumetric Bone Mineral Density at the Radius | 1199.41 (33.69) | 1201.55 (30.10) | 1199.88 (32.70) | 1201.16 (31.10)
  Baseline Total Volumetric Bone Mineral Density at the Tibia: number analyzed (Participants) | 331 | 330 | 336 | 325
  Baseline Total Volumetric Bone Mineral Density at the Tibia | 295.29 (48.05) | 299.23 (49.29) | 297.55 (48.48) | 296.96 (48.94)
  Year 2 Total Volumetric Bone Mineral Density at the Tibia: number analyzed (Participants) | 294 | 284 | 296 | 282
  Year 2 Total Volumetric Bone Mineral Density at the Tibia | 296.76 (49.31) | 303.21 (48.76) | 300.91 (48.88) | 298.90 (49.41)
  Baseline Trabecular Volumetric Bone Mineral Density at the Tibia: number analyzed (Participants) | 331 | 330 | 336 | 325
  Baseline Trabecular Volumetric Bone Mineral Density at the Tibia | 246.63 (40.74) | 250.14 (42.28) | 248.45 (41.14) | 248.31 (41.98)
  Year 2 Trabecular Volumetric Bone Mineral Density at the Tibia: number analyzed (Participants) | 294 | 284 | 296 | 282
  Year 2 Trabecular Volumetric Bone Mineral Density at the Tibia | 249.30 (41.54) | 254.07 (42.02) | 252.11 (41.68) | 251.15 (42.01)
  Baseline Cortical Volumetric Bone Mineral Density at the Tibia: number analyzed (Participants) | 322 | 329 | 333 | 318
  Baseline Cortical Volumetric Bone Mineral Density at the Tibia | 1167.39 (32.26) | 1162.02 (30.38) | 1163.59 (33.09) | 1165.81 (29.56)
  Year 2 Cortical Volumetric Bone Mineral Density at the Tibia: number analyzed (Participants) | 294 | 285 | 298 | 281
  Year 2 Cortical Volumetric Bone Mineral Density at the Tibia | 1169.98 (32.74) | 1166.38 (30.62) | 1166.61 (33.22) | 1169.90 (30.06)

4. Other Pre Specified Outcome: Body Composition
Description: To determine whether vitamin D and/or omega-3 supplementation results in changes in body composition as assessed by DXA: total body fat and lean mass, and fat mass index and lean mass index, regional fat and lean mass and derived ratios.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 388 | 383 | 388 | 383
kg/m^2
  Body Mass Index | 28.29 (5.24) | 28.32 (5.05) | 28.65 (5.15) | 27.96 (5.12)
  Fat Mass Index | 10.26 (4.04) | 10.28 (3.74) | 10.49 (3.98) | 10.05 (3.79)
  Lean Mass Index | 16.46 (2.34) | 16.46 (2.54) | 16.59 (2.42) | 16.33 (2.46)

5. Primary Outcome: Bone Turnover Beta Crosslaps
Description: To determine whether vitamin D and/or omega-3 supplementation reduces bone turnover, assessed biomarkers of bone resorption (beta crosslaps).
Time Frame: 2 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 200 | 200 | 205 | 195
pg/mL
  Baseline beta crosslaps | 0.40 (0.17) | 0.41 (0.19) | 0.41 (0.19) | 0.40 (0.17)
  Year 2 beta crosslaps | 0.40 (0.17) | 0.42 (0.17) | 0.40 (0.17) | 0.41 (0.17)

ADVERSE EVENTS:
Time Frame: Baseline - 2 years
Groups:
- Active Vitamin D/Active Omega-3 Fatty Acids: Received active vitamin D and active omega-3 fatty acids
- Active Vitamin D/Placebo Omega-3 Fatty Acids: Received active vitamin D and placebo omega-3 fatty acids
- Placebo Vitamin D/Active Omega-3 Fatty Acids: Received placebo vitamin D and active omega-3 fatty acids
- Placebo Vitamin D/Placebo Omega-3 Fatty Acids: Received placebo vitamin D and placebo omega-3 fatty acids
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo | Active Vitamin D/Active Omega-3 Fatty Acids | Active Vitamin D/Placebo Omega-3 Fatty Acids | Placebo Vitamin D/Active Omega-3 Fatty Acids | Placebo Vitamin D/Placebo Omega-3 Fatty Acids
All-Cause Mortality (participants affected / at risk) | 8/388 | 3/383 | 3/388 | 8/383 | 2/193 | 6/195 | 1/195 | 2/188
Serious Adverse Events (participants affected / at risk) | 39/388 | 37/383 | 35/388 | 41/383 | 20/193 | 19/195 | 15/195 | 22/188
Other Adverse Events (participants affected / at risk) | 301/388 | 280/383 | 286/388 | 295/383 | 152/193 | 149/195 | 134/195 | 146/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Vitamin D (N=388) | Vitamin D Placebo (N=383) | Active Omega-3 Fatty Acids (N=388) | Omega-3 Fatty Acids Placebo (N=383) | Active Vitamin D/Active Omega-3 Fatty Acids (N=193) | Active Vitamin D/Placebo Omega-3 Fatty Acids (N=195) | Placebo Vitamin D/Active Omega-3 Fatty Acids (N=195) | Placebo Vitamin D/Placebo Omega-3 Fatty Acids (N=188)
Malignant Cancer (General disorders) | 22 | 19 | 15 | 26 | 9 | 13 | 6 | 13
Major Cardiovascular Events (Cardiac disorders) | 7 | 4 | 7 | 4 | 5 | 2 | 2 | 2
Gastrointestinal Bleeding (Gastrointestinal disorders) | 10 | 10 | 9 | 11 | 6 | 4 | 3 | 7
Hypercalcemia (Endocrine disorders) | 3 | 5 | 7 | 1 | 3 | 0 | 4 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Vitamin D (N=388) | Vitamin D Placebo (N=383) | Active Omega-3 Fatty Acids (N=388) | Omega-3 Fatty Acids Placebo (N=383) | Active Vitamin D/Active Omega-3 Fatty Acids (N=193) | Active Vitamin D/Placebo Omega-3 Fatty Acids (N=195) | Placebo Vitamin D/Active Omega-3 Fatty Acids (N=195) | Placebo Vitamin D/Placebo Omega-3 Fatty Acids (N=188)
Kidney Stones (Renal and urinary disorders) | 17 | 11 | 16 | 12 | 10 | 7 | 6 | 5
Parathyroid Condition (Endocrine disorders) | 1 | 4 | 3 | 2 | 0 | 1 | 3 | 1
Kidney Failure or Dialysis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood in Urine (Renal and urinary disorders) | 18 | 27 | 22 | 23 | 8 | 10 | 14 | 13
Easy Bruising (Skin and subcutaneous tissue disorders) | 62 | 61 | 59 | 64 | 29 | 33 | 30 | 31
Frequent Nosebleeds (General disorders) | 10 | 20 | 17 | 13 | 7 | 3 | 10 | 10
Stomach Pain (Gastrointestinal disorders) | 145 | 128 | 139 | 134 | 77 | 68 | 62 | 66
Nausea (Gastrointestinal disorders) | 88 | 77 | 80 | 85 | 43 | 45 | 37 | 40
Constipation (Gastrointestinal disorders) | 121 | 133 | 118 | 136 | 53 | 68 | 65 | 68

LIMITATIONS AND CAVEATS:
Timeline limited to 2 years of follow-up; results not adjusted for multiple hypothesis testing, so findings from the secondary and subgroup analyses are exploratory; results are not generalizable to younger individuals or adults with osteoporosis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT01747447/Prot_SAP_000.pdf